CLINICAL TRIAL: NCT00696046
Title: Direct Intra Bone Marrow Injection Of Unrelated Cord Blood Cells To Improve Engraftment And Reduce Acute Graft-Versus-Host Disease
Brief Title: Intra Bone Marrow Injection Of Unrelated Cord Blood Cells
Acronym: CB01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: francesco frassoni MD, A.O. Universitaria San Martino - Center Stem cells and cell therapy"
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB01-139
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Hematologic Diseases
Keywords: CORD BLOOD CELLS; INTRA BONE MARROW INJECTION; ENGRAFTMENT; transplants
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intrabone Marrow Injection — Cord blood CB units will be thawed in a 37° CB cells will be resuspended in 20ml salinesolution + dextran/albumin, and aliquoted in 4 syringes of 5ml Pts were prepared in a surgical & steril room The anaesthesia consist in a short propofol sedation The injection will last 8-15 minutes. 1° sedation is established, a standard needle for bone marrow aspiration (14 gauge) was inserted few cms in the supero-posterior iliac crest then, an aspiration of about 0.5-1 ml will be performed to assess that the needle was securely introduced in the bone marrow cavity After, we will insert the syringe containing 4-5ml of CB cell suspension which will be gently infused This procedure will be then repeated for all the remaining aliquots at a distance of 2-3cm from the previous one following the iliac crest

SUMMARY:
Compared to other stemcell sources cord blood (CB) is easier and safer to procure, has no donor attrition, a limitless supply, reduced viral transmission, less acute & chronic GVHD, is rich in hematopoietic progenitor cells, and immaturity of T-cell-mediated immunity. CB has delayed neutrophil and platelet engraftment, a prolonged immune reconstitution, uncertain graft-vs-tumor activity, and cell doses from single CB units (U) are a limiting factor for larger recipients Using the intravenous route (IV), a close match between the patient (pts) and the donor or CBU can improve a pts outcome after transplant. Even though a closely matched CBU is preferred, the studies suggest the match may not have to be as close as is needed for marrow or peripheral blood transplants If one has an uncommon tissue type, the doctor may not find a closely matched adult donor and a CBU may be an option, are stored and ready to use. GVHD is a complication after an allogeneic transplant. Studies founded that after a CBtransplant, fewer pts get GVHD than after marrow or peripheral blood transplants. Pts in the studies who did get GVHD after CBtransplant tended to get less severe cases We hypothesized that direct intrabone transplant of CBcells could improve haematologic recovery due to a better stem cell homing, based on the following observations: stem cells recirculate in animals irradiated with limb shielding; a limited fraction (10-15%) of cells injected iv to the haematopoietic sites, possibly because the large majority is lost in other organs; in a mousemodel, HSC directly injected ib repopulated the marrow of lethally irradiated mice 10times more efficiently than HSC cells injected iv; delayed engraftment after CB transplant is possibly not caused by insufficient stem cell numbers; indeed, children grafted with CB cells have superior stem cell reservoir 1year posttransplant when compared to marrow transplant recipients Based on these data, we set-up a phase I-II study to evaluate whether ib injection could be safely performed and whether this procedure could ensure engraftment and shorten the time of complete hematopoietic recovery in adults with high risk haematopoietic malignancies compared to the published data. Neutrophil recovery >80% at day60 and Platelets recovery >80% at days100 were defined as success. 1° endpoint was the probability of neutrophils and platelets recovery after ib CB transplant, 2° included incidence of acute GVHD, relapse, overall survival

DETAILED DESCRIPTION:
Study Design Phase I-II study. Neutrophil recovery > 80% at day 60 and Platelets recovery > 80% at days 100 are defined as success. The limit of 60 days for neutrophil recovery was chosen because it represents the time at which rescue with a second transplant is decided in case of failure to engraft; the day 100 for platelets recovery is taken corresponds to first form reported after transplant to the European Blood and Marrow Transplant Registry.

HLA-A and -B antigens will be identified by low resolution DNA typing, whereas HLA-DRB1 type was determined by high resolution DNA typing techniques. HLA-A, HLA-B, and HLA-DRB1 typing was used to select the most closely matched donor unit-recipient pair, with preference given to HLA-DRB1-matched unit

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematologic malignancies and other forms of hematologic diseases including aplastic anemia
2. Patients will be eligible to enter the study when: A) an unrelated stem cell transplantation was indicated; b) no suitable unrelated HLA-matched donors will be identified in a clinically useful time-frame.
3. Age 16-70
4. Serum creatinine <1.5 mg/dL or Creatinine Clearance >50 ml/min
5. Serum bilirubin <1.5 mg/dl, SGPT <3 x upper limit of normal
6. Negative serology for HIV
7. Central Venous access (Central KT) secured through an indwelling catheter.
8. Life expectancy is not severely limited by concomitant illness.
9. Written and signed informed consent

Exclusion Criteria:

1. Acute Myocardial Infarction (AMI) within the last 12 months
2. Positive pregnancy test
3. Positive HIV serology
4. Chronic renal insufficiency (Serum creatinine >1.5 mg/dl or creatinine cleareance <=50 ml/min)
5. Patient has another progressive malignant disease or a history of other malignancies within 2 years prior to study entry.
6. Severe psychiatric illness or any disorder that compromises ability to give truly informed consent for participation in this study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-12 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
the safety and the probability of neutrophils and platelets recovery after i.b. cord blood transplant. | Full blood count, Monitoring Infections post Transplant, Bone marrow evaluation, Chimerism Analysis, Haematopoietic Reconstitution

SECONDARY OUTCOMES:
the incidence/severity of acute Graft-versus-Host Disease, relapse and overall survival. | Graft-versus-host disease was scored according to current criteria (13).

CONTACTS AND LOCATIONS:
Overall Officials: francesco frassoni, MD, Principal Investigator — A.O. San martino
Locations (1):
- A.O. San Martino - Dep. Center Stem cells and cell therapy", Genoa, genoa, Italy

REFERENCES:
- [Derived] Frassoni F, Gualandi F, Podesta M, Raiola AM, Ibatici A, Piaggio G, Sessarego M, Sessarego N, Gobbi M, Sacchi N, Labopin M, Bacigalupo A. Direct intrabone transplant of unrelated cord-blood cells in acute leukaemia: a phase I/II study. Lancet Oncol. 2008 Sep;9(9):831-9. doi: 10.1016/S1470-2045(08)70180-3. Epub 2008 Aug 8. PMID 18693069